CLINICAL TRIAL: NCT01697865
Title: Reverse Shoulder Arthroplasty With or Without Concomitant Latissimus and Teres Major Transfer for Shoulder Pseudoparalysis With Teres Minor Dysfunction: A Prospective, Randomized Investigation
Brief Title: Reverse Shoulder Arthroplasty With or Without Concomitant Latissimus and Teres Major Transfer for Shoulder Pseudoparalysis With Teres Minor Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 061217B
Record Dates: First submitted 2012-09-27; First posted 2012-10-02 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Osteoarthritis of the Shoulder
Keywords: Reverse total shoulder
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transfer group (Active Comparator): The first surgical technique includes a concomitant latissimus and teres major transfer (transfer group).
  Interventions: Procedure: Transfer group
- Control group (Active Comparator): The second technique does not include a concomitant latissimus and teres major transfer (control group).
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: Transfer group
  Arms: Transfer group
Procedure: Control group
  Arms: Control group

SUMMARY:
The overall objective of this study is to compare the clinical benefit and safety of two different surgical techniques of primary reverse total shoulder arthroplasty for the treatment of shoulder pseudoparalysis from chronic rotator cuff disease with associated teres minor dysfunction. The first surgical technique includes a concomitant latissimus and teres major transfer (transfer group) and the second technique does not include a concomitant latissimus and teres major transfer (control group).

ELIGIBILITY:
Inclusion Criteria:

* Shoulder pseudoparalysis due to chronic rotator cuff dysfunction with or without glenohumeral arthritis.
* Chronic rotator cuff tear with severe retraction, atrophy, fatty infiltration.
* Active forward elevation of less than 90 degrees
* Teres minor dysfunction
* Positive lag and hornblower sign
* Grade 2 or greater fatty infiltration of the teres minor and infraspinatous seen on MRI
* Able to attend scheduled office visits
* Meet all criteria to have a latissimus and teres major transfer

Exclusion Criteria:

* Revision arthroplasty
* Previous shoulder infection
* Neuro-muscular disorder (ie: Parkinson's)
* Advanced dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-06-21 (Actual); Primary Completion 2019-02-12 (Actual); Study Completion 2020-09-21 (Actual)

PRIMARY OUTCOMES:
ADLER Score | 2 Year
  Activities of Daily Living and External Rotation (ADLER) Score: This tool measures patients' ability to do various tasks on a daily basis.

SECONDARY OUTCOMES:
DASH Score | 1 Year, 2 Year
  Disabilities of the Arm, Shoulder, and Hand score
ASES score | 1 Year, 2 Year
  American Shoulder and Elbow Surgeons Score
SF-12 Score | 1 Year, 2 Year
  General Health Outcome score
Range of Motion | 1 Year, 2 Year
  Shoulder range of motion
X-Ray Measurements | 1 Year, 2 Year
  X-ray measurements from the anteroposterior (AP) and axillary views of the shoulder.

CONTACTS AND LOCATIONS:
Locations (1):
- OrthoCarolina Research Institute, Charlotte, North Carolina, United States